CLINICAL TRIAL: NCT01109420
Title: Clinical and Genetic Studies in Familial Non-Medullary Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100102; 10-DK-0102
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-11-19

CONDITIONS: Non-Medullary Thyroid Cancer
Keywords: Hereditary Cancer; Susceptibility Gene(s) for Thyroid Cancer; Screening at Risk Family Members; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/ Cohort 1: Affected with non-medullary thyroid cancer
- 2/ Cohort 2: Non-affected members of families with non-medullary thyroid cancer

SUMMARY:
Background:

- Researchers are studying types of thyroid cancer that seem to cluster in families. Non-medullary thyroid cancer accounts for the vast majority of all types of thyroid cancer, but little is known about possible genes that may cause the cancer. More research is needed to develop the best ways to screen for familial non-medullary thyroid cancer (FNMTC) so that it can be diagnosed and treated at an early stage.

Objectives:

* To evaluate the natural history of FNMTC.
* To determine the best screening strategy for FNMTC.
* To identify genes that may indicate susceptibility to FNMTC.

Eligibility:

- Individuals at least 7 years of age who have two first-degree relatives (e.g., parents, children, siblings) who have or have had non-medullary thyroid cancer or a documented diagnosis of non-medullary thyroid cancer and one living relative with documented non-medullary thyroid cancer.

Design:

* Participants will be evaluated by family history pedigree, physical examination, imaging (including possible neck ultrasound and radioactive iodine scans), and laboratory testing.
* Participants who agree to have blood or other biological samples collected will be asked to enroll in an additional study to provide the appropriate samples and tissues.
* After the initial study evaluation, participants who are not found to have a malignant thyroid tumor will be re-screened every year with non-invasive imaging studies. Participants who are found to have a malignant thyroid tumor will be informed of possible treatment options.

DETAILED DESCRIPTION:
Study Description:

This is a prospective cohort study of individuals with or at risk for non-medullary thyroid cancer. Individuals will be studied over time within the context of their families in order to quantify prospective risks of cancers in family members, to establish the natural history of FNMTC, define the spectrum of diseases within the families, to identify precursor states, to try to assess the contribution of genetic and environmental components of risk, and to develop effective screening strategies.

Objectives:

1. To evaluate the natural history of familial non-medullary thyroid cancer (FNMTC).
2. To determine the best screening strategy for FNMTC.
3. To identify susceptibility gene(s) for FNMTC.

Endpoints:

Not applicable

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will be selected for this protocol based on either a clinical diagnosis of non-medullary thyroid cancer and the presence of one family member with the disease or the presence of 2 living family members with this disease. Patient selection for this protocol will not be based on gender, race, or ethnic background.

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Adults or minor (>= 7 years+), males and females.
* An unaffected individual with (Bullet) 2 first-degree relatives who have or have had nonmedullary thyroid cancer

OR

-An affected individual with documented diagnosis of non-medullary thyroid cancer and (Bullet) one living relative with documented non-medullary thyroid cancer (Note: as this is a familial study, subjects do not need to present with the disease)

OR

* Any member of an affected family. (Note: for this study, an affected family is defined as a family having 2 or more 1st degree relatives with a documented diagnosis of FNMTC.)
* Adults must be able to understand and the willingness to sign the informed consent document.
* Adults must be able to complete the family history questionnaire.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be not be allowed to enroll in this study:

-Subjects unwilling/unable to give informed consent.

Ages: 7 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An individual with 2 first-degree relatives who have or have had non-medullary thyroid cancer or a documented diagnosis of non-medullary thyroid cancer and one living relative with documented non-medullary thyroid cancer (Note: as this is a familial study, subjects do not need to present with the disease) OR Any member of an affected family. (Note: for this study, an affected family is defined as a family having 2 or more 1st degree relatives with a documented diagnosis of FNMTC.)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-08-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the natural history of FNMTC | end of study
  Evaluation the natural history of FNMTC

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Klubo-Gwiezdzinska, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Subject level data will be shared upon request after appropriate collaboration agreements are in place.

REFERENCES:
- [Background] Ito Y, Kakudo K, Hirokawa M, Fukushima M, Yabuta T, Tomoda C, Inoue H, Kihara M, Higashiyama T, Uruno T, Takamura Y, Miya A, Kobayashi K, Matsuzuka F, Miyauchi A. Biological behavior and prognosis of familial papillary thyroid carcinoma. Surgery. 2009 Jan;145(1):100-5. doi: 10.1016/j.surg.2008.08.004. Epub 2008 Sep 21. PMID 19081481
- [Background] Vriens MR, Suh I, Moses W, Kebebew E. Clinical features and genetic predisposition to hereditary nonmedullary thyroid cancer. Thyroid. 2009 Dec;19(12):1343-9. doi: 10.1089/thy.2009.1607. PMID 20001717
- [Background] Chen AY, Jemal A, Ward EM. Increasing incidence of differentiated thyroid cancer in the United States, 1988-2005. Cancer. 2009 Aug 15;115(16):3801-7. doi: 10.1002/cncr.24416. PMID 19598221
- [Background] Chuki E, Behairy N, Auh S, Makarewicz A, Uttarkar Vikram CN, Kumari S, Veeraraghavan P, Cochran C, Gubbi S, Klubo-Gwiezdzinska J. Comparison of Progression-Free Survival in Familial Non-Medullary Thyroid Cancer and Sporadic Differentiated Thyroid Cancer Patients. Thyroid. 2025 Jun;35(6):642-651. doi: 10.1089/thy.2024.0588. Epub 2025 May 20. PMID 40392709
- [Derived] Klubo-Gwiezdzinska J, Yang L, Merkel R, Patel D, Nilubol N, Merino MJ, Skarulis M, Sadowski SM, Kebebew E. Results of Screening in Familial Non-Medullary Thyroid Cancer. Thyroid. 2017 Aug;27(8):1017-1024. doi: 10.1089/thy.2016.0668. Epub 2017 Jul 19. PMID 28657510
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-DK-0102.html